CLINICAL TRIAL: NCT04973631
Title: The Effects of Sex and Age Differences on Gastric Cancer in Terms of Incidence of Histologic Subtypes and Survival Rate: a Retrospective Study
Brief Title: The Effects of Sex and Age Differences on Gastric Cancer : a Retrospective Study
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Nayoung Kim, Professor, Seoul National University Bundang Hospital
Other Study IDs: B-2006-618-004
Record Dates: First submitted 2021-07-13; First posted 2021-07-22 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Sex; Age; Gastric Cancer
MeSH Terms: conditions — Coitus; Stomach Neoplasms | interventions — Sex; Aging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Sex, Age — Evaluate the effect of sex and age on the incidence and survival of GC.

SUMMARY:
Gastric cancer (GC) is more prevalent in males than in females. One of these differences could be the effect of sex hormones such as estrogens. However, few reports have been reported regarding sex and age differences of incidence and survival of GC. The aim of this study was to evaluate the effect of sex and age on the incidence and survival of GC. And we would like to further analyze single GC and synchronous multiple GC, EBV, etc.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Gastric cancer

exclusion criteria:

* Gastric MALTOMA
* Gastric Lymphoma
* Gastrointestinal stromal tumors (GISTs)

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients diagnosed with Gastric cancer at the Seoul National University Bundang Hospital were analyzed retrospectively from May 2003 to February 2020. The data were collected using clinical data warehouses (CDW), and electronic medical records (EMR) were reviewed as needed.
Sampling Method: Probability Sample
Enrollment: 14900 (Actual)
Dates: Start 2003-05 (Actual); Primary Completion 2021-09 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
Survival rate | up to 120 months
  Survival rate of gastric cancer on sex and age
histologic type | about 18 years
  histologic type of gastric cancer on sex and age

REFERENCES:
- [Derived] Song DH, Kim N, Jo HH, Kim S, Choi Y, Oh HJ, Lee HS, Yoon H, Shin CM, Park YS, Lee DH, Kang SH, Park YS, Ahn SH, Suh YS, Park DJ, Kim HH, Kim JW, Kim JW, Lee KW, Chang W, Park JH, Lee YJ, Lee KH, Kim YH, Ahn S, Surh YJ. Analysis of Characteristics and Risk Factors of Patients with Single Gastric Cancer and Synchronous Multiple Gastric Cancer among 14,603 Patients. Gut Liver. 2024 Mar 15;18(2):231-244. doi: 10.5009/gnl220491. Epub 2023 Mar 29. PMID 36987384
- [Derived] Jo HH, Kim N, Oh HJ, Song DH, Choi Y, Park J, Lee J, Yoon H, Shin CM, Park YS, Lee DH, Lee HS, Park YS, Ahn SH, Suh YS, Park DJ, Kim HH, Kim JW, Kim JW, Lee KW, Chang W, Park JH, Lee YJ, Lee KH, Kim YH, Ahn S. The Clinicopathological Features of Mixed Carcinoma in 7,215 Patients with Gastric Cancer in a Tertiary Hospital in South Korea. Gut Liver. 2023 Sep 15;17(5):731-740. doi: 10.5009/gnl220254. Epub 2022 Dec 13. PMID 36510778
- [Derived] Jo HH, Kim N, Jang J, Choi Y, Park J, Park YM, Ahn S, Yoon H, Shin CM, Park YS, Lee DH, Oh HJ, Lee HS, Park YS, Ahn SH, Suh YS, Park DJ, Kim HH, Kim JW, Kim JW, Lee KW, Chang W, Park JH, Lee YJ, Lee KH, Kim YH. Impact of Body Mass Index on Survival Depending on Sex in 14,688 Patients with Gastric Cancer in a Tertiary Hospital in South Korea. Gut Liver. 2023 Mar 15;17(2):243-258. doi: 10.5009/gnl220104. Epub 2022 Nov 1. PMID 36317512